CLINICAL TRIAL: NCT03475602
Title: A Prospective Cohort Study of Membranous Nephropathy-associated Serological Antibody in Prediction of the Prognosis of Idiopathic Membranous Nephropathy
Brief Title: Membranous Nephropathy-associated Serological Antibody Predict the Prognosis of Idiopathic Membranous Nephropathy
Status: Terminated | Type: Observational
Why Stopped: Our center had adopted a new detection method for anti-PLA2R antibodies in all membranous nephropathy patients.
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GDREC2017318H
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-02

CONDITIONS: Idiopathic Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cyclophosphamide: Drug: Cyclophosphamide，CTX Determination of serum concentration of anti PLA2R antibody and anti TSHD7A antibody
  Interventions: Diagnostic Test: PLA2R; Diagnostic Test: TSHD7A
- Cyclosporin: Drug: Cyclosporin Determination of serum concentration of anti PLA2R antibody and anti TSHD7A antibody
  Interventions: Diagnostic Test: PLA2R; Diagnostic Test: TSHD7A

INTERVENTIONS:
Diagnostic Test: PLA2R — Determination of serum concentration of anti PLA2R antibody
Diagnostic Test: TSHD7A — Determination of serum concentration of anti TSHD7A antibody

SUMMARY:
Idiopathic membranous nephropathy (IMN) remains a common cause of the nephrotic syndrome in adults and one of the leading known causes of end-stage renal disease. Identification of circulating autoantigens provide potential biomarkers for diagnosis and therapy of idiopathic membranous nephropathy. M-type phospholipase A2 receptor (PLA2R) and Thrombospondin type-I domain-containing 7A (THSD7A) were identified as the target antigen in membranous nephropathy with high specificity and the concentration of serum anti-PLA2R antibody and anti-TSHD7A antibody were helpful for predicting disease activity. In our prospective cohort study, hospitalized patients diagnosed as IMN are prospectively studied. Circulating anti-PLA2R antibody and anti-THSD7A antibodies were recently screened by using enzyme-linked sorbent assay(ELISA). This study aims to analyse the difference of clinicopathological characteristics for different concentrations of serum anti PLA2R antibody and anti TSHD7A antibody, and analyze the association between baseline concentrations of serum antibody and disease activity. This study also explored the prediction effects of serum antibody concentrations with different types of therapeutic regimen in IMN and compare the curative effects of different types of therapeutic regimen in different serum antibody concentrations.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients who provided informed consent
* (2) Patients who are diagnosed as membranous nephropathy by renal biopsy
* (3) 18 years of age or older, male or female

Exclusion Criteria:

* (1) identification of Secondary factors such as infectious diseases, rheumatic diseases, tumors, drugs and so on
* (2) Previous medicine history of immunosuppressive medication and corticosteroids
* (3) Patients who are not expected to complete 6 months of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Idiopathic Membranous Nephropathy
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Complete Remission | after treatment for 6 months
  Urinary protein excretion<0.3 g/d (uPCR<300 mg/g or <30 mg/mmol), confirmed by two values at least 1 week apart, accompanied by a normal serum albumin concentration, and a normal SCr.
Partial Remission | after treatment for 6 months
  Urinary protein excretion <3.5 g/d (uPCR <3500 mg/g or <350 mg/mmol) and a 50% or greater reduction from peak values;confirmed by two values at least 1 week apart, accompanied by an improvement or normalization of the serum albumin concentration and stable SCr.

SECONDARY OUTCOMES:
estimated Glomerular filtration rate and serum creatinine | after treatment for 6 months
  time to a 50% reduction in baseline estimated Glomerular filtration rate (according to CK-EPI) and to doubling of baseline creatinine

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Dept,Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No